CLINICAL TRIAL: NCT02627196
Title: Barostim Neo® - Baroreflex Activation Therapy® for Heart Failure
Brief Title: Baroreflex Activation Therapy for Heart Failure
Acronym: BeAT-HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CVRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 360043-001
Record Dates: First submitted 2015-12-07; First posted 2015-12-10 (Estimated); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Practice Management, Medical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Device and Medical Management (Experimental): Subjects will be implanted with the BAROSTIM NEO System and receive optimal, stable, Guideline Directed Medical Therapy (GDMT) for heart failure (American Heart Association [AHA] / American College of Cardiology [ACC] guidelines), including drugs to be determined by the subject's physician. Drug types include: Loop Diuretics, Thiazide Diuretics, Potassium-sparing Diuretics, Sequential Nephron Blockade, ACE Inhibitors, ARBs, ARNI, Aldosterone Antagonists, Beta Blockers and Hydralazine and Isosorbide Dinitrate.
  Interventions: Device: BAROSTIM NEO® System; Drug: Medical Management
- Medical Management (Active Comparator): Subjects will receive optimal, stable, Guideline Directed Medical Therapy (GDMT) for heart failure (American Heart Association [AHA] / American College of Cardiology [ACC] guidelines), including drugs to be determined by the subject's physician. Drug types include: Loop Diuretics, Thiazide Diuretics, Potassium-sparing Diuretics, Sequential Nephron Blockade, ACE Inhibitors, ARBs, ARNI, Aldosterone Antagonists, Beta Blockers and Hydralazine and Isosorbide Dinitrate.
  Interventions: Drug: Medical Management

INTERVENTIONS:
Device: BAROSTIM NEO® System
  Arms: Device and Medical Management
Drug: Medical Management

SUMMARY:
The purpose of this clinical trial (NCT02627196) is to develop valid scientific evidence for safety and effectiveness of Baroreflex Activation Therapy with the BAROSTIM NEO System in subjects with heart failure, defined as New York Heart Association (NYHA) functional Class III, left ventricular ejection fraction (LVEF) ≤ 35% and NT-proBNP<1600 pg/ml despite being treated with the appropriate heart failure guideline directed therapy, excluding subjects eligible for or actively receiving Cardiac Resynchronization Therapy (CRT).

The total trial duration is anticipated to be approximately 5 years; however, the duration of an individual subject enrollment will depend on when he or she entered the trial.

DETAILED DESCRIPTION:
The BAROSTIM NEO - Baroreflex Activation Therapy for Heart Failure is a prospective, randomized trial in subjects with reduced ejection fraction heart failure. Subjects will be randomized in a 1:1 ratio to receive Barostim Activation Therapy with an implanted BAROSTIM NEO System in addition to medical management or to receive medical management alone (no device implant). The trial will be conducted at up to 120 investigational centers in the U.S. and up to 20 investigational centers outside the U.S. These centers will enroll up to 1200 subjects to randomize approximately 480 subjects who meet the entry criteria.

For all subjects, trial visits will occur at 0.5, 1, 1.5, 2, 3, 6, 9 and 12 months post-implant (post anticipated implant for medical management). Visits will occur quarterly from 15 to 24 months and semi-annually thereafter.

Subjects are followed in an identical manner regardless of trial arm.

The data will provide evidence of the safety and efficacy of BAROSTIM THERAPY. The accumulated morbidity and mortality data collected will provide evidence of morbidity and mortality benefit. This trial will involve one or more interim analyses to evaluate when sufficient evidence is reached for the final morbidity and mortality analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 years or above.
2. Currently NYHA Class II or III heart failure. For NYHA Class II, must have been NYHA Class III at any point in time within 3 calendar months prior to enrollment or at time of screening (enrollment is defined as the date the subject provided written consent).
3. Left ventricular ejection fraction ≤ 35% within 45 days prior to randomization.
4. Heart failure accompanied by either:

   * Core lab NT-proBNP ≥ 400 AND <1600 pg/ml within 45 days prior to randomization OR
   * Core lab NT-proBNP < 400 pg/ml within 45 days prior to randomization AND a heart failure hospitalization in the past 12 months.

   Note: Heart failure hospitalization may include an overnight hospital or hospital-based observation unit stay with a primary diagnosis of heart failure or an emergency room visit with a primary diagnosis of heart failure.

   Note: Screening/Baseline core lab NT-proBNP must be collected in an outpatient setting at a time when the subject is thought to be clinically stable.
5. On optimal, stable, Guideline Directed Medical Therapy (GDMT) per country specific guidelines for the treatment of heart-failure throughout screening/baseline evaluation and for at least 4 weeks prior to obtaining any post-consent screening parameters:

   * No more than a 100% increase or a 50% decrease of the dosage of any one medication other than a diuretic.
   * Medication changes within a drug class are allowed as long as the equivalent dosage is within the limits specified above.
   * Unrestricted changes in diuretics are allowed as long as the subject remains on a diuretic.
6. Six-minute hall walk (6MHW) ≥ 150 m AND ≤ 400 m within 45 days prior to randomization.
7. The artery planned for the BAROSTIM implant must meet both of the following criteria:

   * At least one carotid bifurcation as identification by a bilateral carotid duplex ultrasound within 6 months prior to randomization that is:

     1. Below the level of the mandible AND
     2. No ulcerative carotid arterial plaques AND
     3. No carotid atherosclerosis producing a 50% or greater reduction in linear diameter in the internal carotid AND
     4. No carotid atherosclerosis producing a 50% or greater reduction in linear diameter in the distal common carotid
   * No prior surgery, radiation, or endovascular stent placement in the carotid artery or the carotid sinus region.
8. If female and of childbearing potential, must use a medically accepted method of birth control (e.g., barrier method with spermicide, oral contraceptive, or abstinence) and agree to continue use of this method for the duration of the trial. Women of childbearing potential must have a negative pregnancy test within 14 days prior to randomization.
9. Received a standard cardiac work up and is an appropriate candidate for the study and the surgical procedure as determined by a trial cardiologist and a trial surgeon.
10. Subjects implanted with a cardiac rhythm management device that does not utilize an intracardiac lead, or implanted with a neurostimulation device, must be approved by the CVRx Clinical department.
11. Signed a CVRx-approved informed consent form for participation in this trial.

Exclusion Criteria:

If any of the following criteria are met, subjects are not eligible for this trial.

1. Received cardiac resynchronization therapy (CRT) within six months of randomization, or is actively receiving CRT.
2. Currently have a Class I indication for a cardiac resynchronization therapy (CRT) device according to AHA/ACC/ESC guidelines for the treatment of congestive heart failure. ,
3. Known or suspected baroreflex failure or autonomic neuropathy.
4. AHA/ACC Stage D heart failure within 45 days prior to randomization.
5. Body mass index > 40.
6. Serum estimated glomerular filtration rate (eGFR) < 25 mL/min/1.73 m2 within 45 days prior to randomization.
7. Recurring resting heart rate of either < 60 bpm or > 100 bpm via clinic measurements within 45 days prior to randomization. (Note: Heart rate <60 bpm is not applicable to subjects with an implanted device capable of pacing.)
8. Recurring symptomatic hypotension within 45 days prior to randomization.
9. Significant uncontrolled symptomatic bradyarrhythmias or unstable ventricular arrhythmias.
10. Subjects with any surgery that has occurred, or is planned to occur, within 45 days of the BAROSTIM NEO implant procedure. This includes pacemaker or ICD implants or battery replacements.
11. Episode of NYHA class IV heart failure with acute pulmonary edema within 45 days prior to randomization.
12. Any of the following within 3 months of randomization:

    * Myocardial infarction
    * Unstable angina
    * Percutaneous coronary intervention (e.g. CABG or PTCA)
    * Cerebral vascular accident or transient ischemic attack
    * Sudden cardiac death
13. Solid organ or hematologic transplant, or currently being actively evaluated for an organ transplant.
14. Has received or is receiving LVAD therapy.
15. Has received or is receiving chronic dialysis.
16. Heart failure secondary to a reversible cause, such as cardiac structural valvular disease, acute myocarditis and pericardial constriction.
17. Primary pulmonary hypertension.
18. Infiltrative cardiomyopathy (e.g. cardiac amyloidosis).
19. Severe COPD or severe restrictive lung disease (e.g. requires chronic steroid use or home oxygen use).
20. Active malignancy.
21. Current or planned treatment with intravenous positive inotrope therapy.
22. Life expectancy less than one year.
23. Clinically significant psychological condition that in the physician's opinion would prohibit the subject's ability to meet the protocol requirements.
24. Unable or unwilling to fulfill the protocol medication compliance, testing, and follow-up requirements (e.g. recent drug abuse).
25. Enrolled and active in another (e.g. device, pharmaceutical, or biological) clinical trial unless approved by the CVRx Clinical department.
26. Subjects with known allergies to silicone and titanium.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2016-04-19 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Cardiovascular Mortality and Heart Failure Morbidity | At study completion, approximately 5 years
  To demonstrate that treatment with the BAROSTIM NEO® System, relative to medical management, reduces the rate of cardiovascular mortality or worsening heart failure that leads to hospitalization, cardiac assist device or heart transplant.
Major Adverse Neurological and Cardiovascular Events (MANCE) | 6 months post implant
  To demonstrate the safety of the Barostim NEO® System via the event-free rate of all system- and procedure-related Major Adverse Neurological and Cardiovascular Events (MANCE) occurring within 6 months post implant in the device arm.
Amino-terminal prohormone of brain natriuretic peptide (NT-proBNP) | 6 months post implant
  To demonstrate that treatment with the BAROSTIM NEO® system results in a larger reduction in NT-proBNP at 6 months than medical management.
Six Minute Hall Walk (6MHW) | 6 months post implant.
  To demonstrate that treatment with the BAROSTIM NEO® system results in a larger improvement in 6MHW at 6 months than medical management
Minnesota Living With Heart Failure Quality of Life (MLWHF QOL) | 6 months post implant
  To demonstrate that treatment with the BAROSTIM NEO® System results in a larger improvement in MLWHF QOL at 6 months than medical management

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zile, MD, Study Chair — Medical University of South Carolina; William Abraham, MD, Principal Investigator — Ohio State University; Fred Weaver, MD, Principal Investigator — University of Southern California; Faiez Zannad, MD, Principal Investigator — Inserm Centre d'Investigation, CHU de Nancy; JoAnn Lindenfield, MD, Principal Investigator — Vanderbilt Heart and Vascular Institute
Locations (92):
- United States (88):
  - Heart and Rhythm Solutions, PLLC, Chandler, Arizona
  - Chan Heart Rhythm Institute, Mesa, Arizona
  - Arizona Arrhythmia Research Center, Phoenix, Arizona
  - Phoenix Cardiovascular Research Group, Phoenix, Arizona
  - Cardiovascular Consultants, Ltd., Phoenix, Arizona
  - Washington Regional Medical Center, Fayetteville, Arkansas
  - Central Cardiology Medical Center, Bakersfield, California
  - Chula Vista Cardiac Center, Chula Vista, California
  - Sharp Grossmont, Chula Vista, California
  - Sharp Chula Vista Medical Center, Chula Vista, California
  - John Muir Health Clinical Research Center, Concord, California
  - University of California, San Francisco - Fresno, Fresno, California
  - Herndon Surgery Center, Fresno, California
  - Glendale Adventist Medical Center, Glendale, California
  - Memorial Health Services, Laguna Hills, California
  - Los Alamitos Cardiovascular, Los Alamitos, California
  - Southern California Permanente Medical Group, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - Advanced Cardiovascular Specialists, Mountain View, California
  - Hoag Memorial Hospital, Newport Beach, California
  - UC Irvine Health, Orange, California
  - Desert Heart Regional Medical Center, Palm Springs, California
  - Huntington Hospital, Pasadena, California
  - Dignity Health, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - Bonometti, Inc, Santa Barbara, California
  - Adventist Heart Institute, St. Helena, California
  - North Colorado Medical Center, Greeley, Colorado
  - Medical Center of the Rockies Research, Loveland, Colorado
  - Atlantic Clinical Research Center - Cardiology, Atlantis, Florida
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Memorial Cardiovascular Institute, Hollywood, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Avanza Medical Research Center, Pensacola, Florida
  - University of South Florida, Tampa, Florida
  - Mercer University, Macon, Georgia
  - WellStar Medical Group, Marietta, Georgia
  - St. Alphonsus Medical Center, Boise, Idaho
  - NorthShore University Health System, Evanston, Illinois
  - Advocate Medical Group, Naperville, Illinois
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - Via Christi Research, Wichita, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Tulane University & Vascular Institute, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - St. Elizabeth's Medical Center, Brighton, Massachusetts
  - Detroit Medical Center Cardiovascular Institute, Detroit, Michigan
  - Ascension St. Mary's Research Institute, Saginaw, Michigan
  - Providence-Providence Park Hospital, Southfield, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mercy Hospital Springfield, Springfield, Missouri
  - Washington University, St Louis, Missouri
  - St. Louis Heart and Vascular, St Louis, Missouri
  - Mercy Hospital St. Louis, St Louis, Missouri
  - Nebraska Heart Institute, Lincoln, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Healthcare Partners Clinical Research, Las Vegas, Nevada
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Presbyterian Heart Group, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - St. Francis Hospital - Long Island, Roslyn, New York
  - Cone Health, Greensboro, North Carolina
  - WakeMed, Raleigh, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Oklahoma Cardiovascular Research Group, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Drexel University, Philadelphia, Pennsylvania
  - Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - McLeod Cardiology Associates, Florence, South Carolina
  - Stern Cardiovascular Foundation, Germantown, Tennessee
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Cardiovascular Research Institute of Dallas, Dallas, Texas
  - Private Practice Leadership, Houston, Texas
  - Methodist Richardson Medical Center, Richardson, Texas
  - Tyler Cardiovascular Consultants, Tyler, Texas
  - Intermountain Heart Institute, Murray, Utah
  - University of Utah, Salt Lake City, Utah
  - Virginia Mason Medical Center, Seattle, Washington
  - CHI Franciscan Health Research Center, Tacoma, Washington
  - Columbia St. Mary's Hospital, Milwaukee, Wisconsin
- United Kingdom (4):
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge, Cambridgeshire
  - Liverpool Heart and Chest Hospital, Liverpool, Merseyside
  - Royal Brompton & Harefield NHS Foundation Trust, Harefield, Middlesex
  - Belfast Health & Social Care Trust, Belfast, Northern Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fu Q, Zhang R, Witkowski S, Arbab-Zadeh A, Prasad A, Okazaki K, Levine BD. Persistent sympathetic activation during chronic antihypertensive therapy: a potential mechanism for long term morbidity? Hypertension. 2005 Apr;45(4):513-21. doi: 10.1161/01.HYP.0000158312.63381.c1. Epub 2005 Feb 28. PMID 15738344
- [Background] Esler M, Kaye D. Increased sympathetic nervous system activity and its therapeutic reduction in arterial hypertension, portal hypertension and heart failure. J Auton Nerv Syst. 1998 Oct 15;72(2-3):210-9. doi: 10.1016/s0165-1838(98)00107-6. PMID 9851571
- [Background] Sleight P. The importance of the autonomic nervous system in health and disease. Aust N Z J Med. 1997 Aug;27(4):467-73. doi: 10.1111/j.1445-5994.1997.tb02220.x. PMID 9448899
- [Background] Peters TK, Koralewski HE, Zerbst E. Blood pressure and heart rate changes during physical activity upon heart rate feedback-controlled electrical carotid sinus nerve stimulation. Int J Cardiol. 1989 Mar;22(3):389-92. doi: 10.1016/0167-5273(89)90281-7. PMID 2785088
- [Background] Georgakopoulos D, Wagner D, Cates AW, Irwin E, Lovett EG. Effects of electrical stimulation of the carotid sinus baroreflex using the Rheos device on ventricular-vascular coupling and myocardial efficiency assessed by pressure-volume relations in non-vagotomized anesthetized dogs. Annu Int Conf IEEE Eng Med Biol Soc. 2009;2009:2025-9. doi: 10.1109/IEMBS.2009.5334421. PMID 19964769
- [Background] Sabbah HN, Gupta RC, Imai M, Irwin ED, Rastogi S, Rossing MA, Kieval RS. Chronic electrical stimulation of the carotid sinus baroreflex improves left ventricular function and promotes reversal of ventricular remodeling in dogs with advanced heart failure. Circ Heart Fail. 2011 Jan;4(1):65-70. doi: 10.1161/CIRCHEARTFAILURE.110.955013. Epub 2010 Nov 19. PMID 21097604
- [Background] Zucker IH, Hackley JF, Cornish KG, Hiser BA, Anderson NR, Kieval R, Irwin ED, Serdar DJ, Peuler JD, Rossing MA. Chronic baroreceptor activation enhances survival in dogs with pacing-induced heart failure. Hypertension. 2007 Nov;50(5):904-10. doi: 10.1161/HYPERTENSIONAHA.107.095216. Epub 2007 Sep 10. PMID 17846349
- [Background] Zile MR, Abraham WT, Weaver FA, Butter C, Ducharme A, Halbach M, Klug D, Lovett EG, Muller-Ehmsen J, Schafer JE, Senni M, Swarup V, Wachter R, Little WC. Baroreflex activation therapy for the treatment of heart failure with a reduced ejection fraction: safety and efficacy in patients with and without cardiac resynchronization therapy. Eur J Heart Fail. 2015 Oct;17(10):1066-74. doi: 10.1002/ejhf.299. Epub 2015 Jun 10. PMID 26011593
- [Background] Weaver FA, Abraham WT, Little WC, Butter C, Ducharme A, Halbach M, Klug D, Lovett EG, Madershahian N, Muller-Ehmsen J, Schafer JE, Senni M, Swarup V, Wachter R, Zile MR. Surgical Experience and Long-term Results of Baroreflex Activation Therapy for Heart Failure With Reduced Ejection Fraction. Semin Thorac Cardiovasc Surg. 2016 Summer;28(2):320-328. doi: 10.1053/j.semtcvs.2016.04.017. Epub 2016 Jun 2. PMID 28043438
- [Background] Ferreira JP, Duarte K, Graves TL, Zile MR, Abraham WT, Weaver FA, Lindenfeld J, Zannad F. Natriuretic Peptides, 6-Min Walk Test, and Quality-of-Life Questionnaires as Clinically Meaningful Endpoints in HF Trials. J Am Coll Cardiol. 2016 Dec 20;68(24):2690-2707. doi: 10.1016/j.jacc.2016.09.936. PMID 27978953
- [Background] Abraham WT, Zile MR, Weaver FA, Butter C, Ducharme A, Halbach M, Klug D, Lovett EG, Muller-Ehmsen J, Schafer JE, Senni M, Swarup V, Wachter R, Little WC. Baroreflex Activation Therapy for the Treatment of Heart Failure With a Reduced Ejection Fraction. JACC Heart Fail. 2015 Jun;3(6):487-496. doi: 10.1016/j.jchf.2015.02.006. Epub 2015 May 14. PMID 25982108
- [Background] Gronda E, Francis D, Zannad F, Hamm C, Brugada J, Vanoli E. Baroreflex activation therapy: a new approach to the management of advanced heart failure with reduced ejection fraction. J Cardiovasc Med (Hagerstown). 2017 Sep;18(9):641-649. doi: 10.2459/JCM.0000000000000544. PMID 28737621
- [Background] Gronda E, Seravalle G, Brambilla G, Costantino G, Casini A, Alsheraei A, Lovett EG, Mancia G, Grassi G. Chronic baroreflex activation effects on sympathetic nerve traffic, baroreflex function, and cardiac haemodynamics in heart failure: a proof-of-concept study. Eur J Heart Fail. 2014 Sep;16(9):977-83. doi: 10.1002/ejhf.138. Epub 2014 Jul 28. PMID 25067799
- [Background] Zile MR, Claggett BL, Prescott MF, McMurray JJ, Packer M, Rouleau JL, Swedberg K, Desai AS, Gong J, Shi VC, Solomon SD. Prognostic Implications of Changes in N-Terminal Pro-B-Type Natriuretic Peptide in Patients With Heart Failure. J Am Coll Cardiol. 2016 Dec 6;68(22):2425-2436. doi: 10.1016/j.jacc.2016.09.931. PMID 27908347
- [Background] Cleland JG, McMurray JJ, Kjekshus J, Cornel JH, Dunselman P, Fonseca C, Hjalmarson A, Korewicki J, Lindberg M, Ranjith N, van Veldhuisen DJ, Waagstein F, Wedel H, Wikstrand J; CORONA Study Group. Plasma concentration of amino-terminal pro-brain natriuretic peptide in chronic heart failure: prediction of cardiovascular events and interaction with the effects of rosuvastatin: a report from CORONA (Controlled Rosuvastatin Multinational Trial in Heart Failure). J Am Coll Cardiol. 2009 Nov 10;54(20):1850-9. doi: 10.1016/j.jacc.2009.06.041. PMID 19892235
- [Background] Anand IS, Rector TS, Cleland JG, Kuskowski M, McKelvie RS, Persson H, McMurray JJ, Zile MR, Komajda M, Massie BM, Carson PE. Prognostic value of baseline plasma amino-terminal pro-brain natriuretic peptide and its interactions with irbesartan treatment effects in patients with heart failure and preserved ejection fraction: findings from the I-PRESERVE trial. Circ Heart Fail. 2011 Sep;4(5):569-77. doi: 10.1161/CIRCHEARTFAILURE.111.962654. Epub 2011 Jun 29. PMID 21715583
- [Background] Anand IS, Claggett B, Liu J, Shah AM, Rector TS, Shah SJ, Desai AS, O'Meara E, Fleg JL, Pfeffer MA, Pitt B, Solomon SD. Interaction Between Spironolactone and Natriuretic Peptides in Patients With Heart Failure and Preserved Ejection Fraction: From the TOPCAT Trial. JACC Heart Fail. 2017 Apr;5(4):241-252. doi: 10.1016/j.jchf.2016.11.015. PMID 28359411
- [Background] Fruhwald FM, Fahrleitner-Pammer A, Berger R, Leyva F, Freemantle N, Erdmann E, Gras D, Kappenberger L, Tavazzi L, Daubert JC, Cleland JG. Early and sustained effects of cardiac resynchronization therapy on N-terminal pro-B-type natriuretic peptide in patients with moderate to severe heart failure and cardiac dyssynchrony. Eur Heart J. 2007 Jul;28(13):1592-7. doi: 10.1093/eurheartj/ehl505. Epub 2007 Feb 13. PMID 17298973
- [Background] Zile MR, Abraham WT, Lindenfeld J, Weaver FA, Zannad F, Graves T, Rogers T, Galle EG. First granted example of novel FDA trial design under Expedited Access Pathway for premarket approval: BeAT-HF. Am Heart J. 2018 Oct;204:139-150. doi: 10.1016/j.ahj.2018.07.011. Epub 2018 Jul 22. PMID 30118942
- [Derived] Lindenfeld J, Gupta R, Grazette L, Ruddy JM, Tsao L, Galle E, Rogers T, Sears S, Zannad F. Response by Sex in Patient-Centered Outcomes With Baroreflex Activation Therapy in Systolic Heart Failure. JACC Heart Fail. 2021 Jun;9(6):430-438. doi: 10.1016/j.jchf.2021.01.012. Epub 2021 May 12. PMID 33992562
- [Derived] Zile MR, Lindenfeld J, Weaver FA, Zannad F, Galle E, Rogers T, Abraham WT. Baroreflex Activation Therapy in Patients With Heart Failure With Reduced Ejection Fraction. J Am Coll Cardiol. 2020 Jul 7;76(1):1-13. doi: 10.1016/j.jacc.2020.05.015. PMID 32616150
- See also: Sponsor Website — http://www.cvrx.com
- See also: Study Website — https://www.beathf.com/